CLINICAL TRIAL: NCT05993871
Title: Diabetic Small Fiber Neuropathy: Clinical, Electrophysiological and Neurosonographic Study
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Sami Alkotami, Assistant Lecturer of Neurology, Tanta University
Other Study IDs: 34059/8/20
Record Dates: First submitted 2023-05-21; First posted 2023-08-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Small Fiber Neuropathy; Diabetic Neuropathies; Autonomic Neuropathy; Diabetic Peripheral Neuropathy; Painful Diabetic Neuropathy; Diabetic Polyneuropathy
MeSH Terms: conditions — Small Fiber Neuropathy; Diabetic Neuropathies | interventions — Physical Examination; Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Distal leg 3mm punch skin biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with diabetic small fiber neuropathy: Diabetic Patients presented with pure small fiber neuropathy.
  Interventions: Diagnostic Test: Clinical Evaluation/Questionnaires; Diagnostic Test: Nerve Conduction Study; Diagnostic Test: Small fiber electrodiagnostic tests; Diagnostic Test: Nerve Ultrasound; Diagnostic Test: Skin Biopsy
- Patients with diabetic mixed small and large fiber neuropathy: Diabetic Patients presented with mixed small and large fiber neuropathy
  Interventions: Diagnostic Test: Clinical Evaluation/Questionnaires; Diagnostic Test: Nerve Conduction Study; Diagnostic Test: Small fiber electrodiagnostic tests; Diagnostic Test: Nerve Ultrasound; Diagnostic Test: Skin Biopsy
- Subjects without neuropathy: Healthy subjects without any symptoms and/or signs suggesting neuropathy, and within average IENFD on skin biopsy.
  Interventions: Diagnostic Test: Clinical Evaluation/Questionnaires; Diagnostic Test: Nerve Conduction Study; Diagnostic Test: Small fiber electrodiagnostic tests; Diagnostic Test: Nerve Ultrasound; Diagnostic Test: Skin Biopsy

INTERVENTIONS:
Diagnostic Test: Clinical Evaluation/Questionnaires — Anthropometric measures, somatosensory assessment (NPS, UENS, TCNS), autonomic assessment (COMPASS-31, Ewing battery), and severity and quality of life evaluation (NPS, TCNS, COMPASS-31, and EuroQOL-5D-5L index score)
Diagnostic Test: Nerve Conduction Study — Routine Nerve Conduction Study.
Diagnostic Test: Small fiber electrodiagnostic tests — R-R interval analysis, Cutaneous Silent Period and Sympathetic Skin Response.
Diagnostic Test: Nerve Ultrasound — Bilateral vagal, left median, right ulnar, left tibial and right sural nerves ultrasound.
Diagnostic Test: Skin Biopsy — distal leg 3mm punch skin biopsy

SUMMARY:
The aim of work is to study the clinical, electrodiagnostic and neurosonographic characteristics of diabetic patients with small fiber neuropathy in the Egyptian population, and to evaluate both the diagnostic and the prognostic impact of the studied factors on the neuropathy severity and quality of life.

DETAILED DESCRIPTION:
This case-control observational study is aiming to evaluate patients with diabetic small fiber neuropathy in the Egyptian.

Diabetic small fiber neuropathy was defined as both of the following:

A. Typical clinical symptoms of SFN such as burning or sharp pain in toes and feet, and on clinical examination: loss of small fiber modalities (pinprick and temperature), hyperalgesia, allodynia, and/or autonomic signs.

B. Reduced intraepidermal nerve fiber density (IENFD) in distal leg skin punch biopsy.

The study includes 3 groups:

Group I: Patients with diabetic small fiber neuropathy Group II (Control Group): Patients with diabetic mixed small and large fiber neuropathy Group III (Control Group): Subjects without peripheral neuropathy

Clinical evaluation includes: Neuropathic Pain 4 (DN4) questionnaire, 11-point Numeric Pain Scale (NPS), Utah Early Neuropathy Scale (UENS), Toronto Clinical Neuropathy Scale (TCNS), Composite Autonomic Symptom Score (COMPASS-31), an Arabic version, and several anthropometric measures; including: body weight in kilograms, height in centimeters, waist circumference measured in centimeters at the top of the iliac crest, and systolic "SBP" and diastolic "DBP" blood pressure measurement in mmHg.

Electrodiagnostic evaluation includes: routine nerve conduction study, cutaneous silent period by stimulating left median nerve and right sural nerve and recording from the abductor pollicis brevis and tibialis anterior muscles, respectively, bilateral hand-to hand and foot-to-foot sympathetic skin response, and Ewing battery using R-R interval analysis, in addition to the blood pressure tests.

Neurosonographic evaluation includes: bilateral vagal nerve scan at the mid-neck lateral to the thyroid cartilage, left median and right ulnar nerves scan at the mid-forearm, left tibial nerve at the distal ankle 2 to 4 fingerbreadths proximal to the medial malleolus, and right sural nerve 2 to 4 fingerbreadths proximal to the lateral malleolus. Nerves are evaluated for transverse cross-sectional area (CSA).

Severity and outcome measures are assessed using: NPS, TCNS, COMPASS-31, and the index score of Euro Quality of Life -5 Dimensions -5 Levels (EuroQOL-5D-5L), the Arabic version.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with diabetes mellitus or impaired glucose intolerance by laboratory investigations including any of the following: HbA1C, fasting blood sugar and 2-hour post prandial blood sugar, and/or antidiabetic medication.
2. Patients presented with small fiber neuropathy (SFN), including all the following:

   A. Typical clinical symptoms of SFN such as burning or sharp pain in toes and feet, and on clinical examination: loss of small fiber modalities (pinprick and temperature), hyperalgesia, allodynia, and/or autonomic signs.

   B. Reduced intraepidermal nerve fiber density (IENFD) in distal leg skin punch biopsy.
3. Age older than 18 years old

Exclusion Criteria:

1. Mental illness that made interviewing ineffective
2. Physical illness leading to language and/or cognitive barrier
3. Other conditions that could cause neuropathy (e.g., chemotherapy, alcohol intake, established vitamin B12 deficiency, established hereditary neuropathy "or first-degree family members", active malignancy, chronic advanced liver or kidney diseases thought to cause neuropathy and history of bariatric surgery).
4. Atrial Fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group I: Patients with diabetic small fiber neuropathy Group II: Patients with diabetic mixed small and large fiber neuropathy Group III: Subjects without neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Demonstrate the findings of UENS in the studied groups | through study completion, an average of 9 months
  Demonstrate the findings of Utah early neuropathy scale in the studied groups to screen for neuropathic symptoms, where overall scores of 4 and more are considered positive.
Demonstrate the findings of TCNS in the studied groups | through study completion, an average of 9 months
  Demonstrate the findings of Toronto clinical neuropathy scale in the studied groups, to screen for the neuropathic symptoms where overall scores of 6 and more are considered positive.
Demonstrate the findings of EuroQOL-5D-5L in the studied groups | through study completion, an average of 9 months
  Demonstrate the findings of Euro quality of life -5 dimensions -5 levels scale in the studied groups, where lesser scores suggest a lower overall quality of life.
Demonstrate the findings of nerve conduction studies protocol of the performed nerves in the studied groups. | through study completion, an average of 9 months
  Demonstrate the findings of nerve conduction studies (NCS) to define neuropathy in the studied groups, which include: unilateral sensory studies of sural, superficial peroneal and ulnar nerves, and motor studies of tibial, peroneal, and ulnar motor nerves with ulnar and tibial F wave latencies. Nerves were evaluated according to a recommended protocol for NCS postulated by the American Academy of Neurology in conjunction with the American Association of Electrodiagnostic Medicine and the American Academy of Physical Medicine and Rehabilitation, which include an abnormality of any nerve conduction attribute is in two separate nerves, one of which must be the sural nerve.
Demonstrate the findings of cutaneous silent period in the studied groups. | through study completion, an average of 9 months
  Demonstrate the findings of cutaneous silent period on stimulating left median nerve and recording from the left abductor pollicis brevis muscle, and on stimulating right sural nerve and recording from the tibialis anterior muscle, where abnormal results in encountered when there is delayed onset and/or end latencies, and/or decreased or absent duration.
Demonstrate the findings of sympathetic skin response in the studied groups. | through study completion, an average of 9 months
  Demonstrate the findings of sympathetic skin response on hand-to-hand stimulation of both median nerves, and foot-to-foot stimulation of both tibial nerves, where abnormal result is encountered when there is absent response, or delayed onset latency and/or decreased amplitude.
Demonstrate the findings of Ewing battery in the studied groups. | through study completion, an average of 9 months
  Demonstrate the findings of Ewing battery in the studied groups, where findings are recorded in all the 5 domains of the battery as normal or borderline or abnormal. Total score ranges from 0-5, and cardiovascular autonomic neuropathy is diagnosed according to the findings o fthe battery, where the findings are classified as follows
  * Normal: If all tests are normal, or one test is borderline.
  * Early: One heart rate test is abnormal or two are borderline.
  * Definite: At least two heart rate tests are abnormal
  * Severe: At least two heart rate tests are abnormal plus either at least one blood pressure test is abnormal or both tests are borderline.
  * Atypical: Any other undefined combination.
  Further simplified classification is either normal (including normal or early findings) and abnormal (including definite, severe and atypical findings).
Demonstrate the findings of nerve ultrasound CSA of both vagal nerves. | through study completion, an average of 9 months
  Demonstrate the findings of nerve ultrasound cross-sectional area of both vagal nerves scanned opposite to the cricoid cartilage in the studied groups.
Demonstrate the findings of nerve ultrasound CSA of right sural nerve. | through study completion, an average of 9 months
  Demonstrate the findings of nerve ultrasound cross-sectional area of right sural nerve at the distal calf in the studied groups.
Demonstrate the findings of nerve ultrasound CSA of left tibial nerve. | through study completion, an average of 9 months
  Demonstrate the findings of nerve ultrasound cross-sectional area of left tibial nerve at the distal calf in the studied groups.
Demonstrate the findings of nerve ultrasound CSA of left median nerve. | through study completion, an average of 9 months
  Demonstrate the findings of nerve ultrasound cross-sectional area of left median nerve at the mid-forearm in the studied groups.
Demonstrate the findings of nerve ultrasound CSA of right ulnar nerve. | through study completion, an average of 9 months
  Demonstrate the findings of nerve ultrasound cross-sectional area of right ulnar nerve at the mid-forearm in the studied groups.

SECONDARY OUTCOMES:
Diabetic neuropathy severity assessment using NPS | through study completion, an average of 9 months
  Diabetic neuropathy severity assessment using 11-item Numeric Pain Scale overall score.
Diabetic neuropathy severity assessment TCNS | through study completion, an average of 9 months
  Diabetic neuropathy severity assessment using Toronto clinical neuropathy scale, overall score.
Diabetic neuropathy severity assessment using COMPASS-31 | through study completion, an average of 9 months
  Diabetic neuropathy severity assessment using The Composite Autonomic Symptom Score-31, overall score.
Diabetic neuropathy quality of life evaluation using Euro quality of life -5 dimensions -5 levels scale. | through study completion, an average of 9 months.
  Diabetic neuropathy quality of life evaluation using EuroQOL-5D-5L index value.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Sami Mahmoud Alkotami, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Devigili G, Tugnoli V, Penza P, Camozzi F, Lombardi R, Melli G, Broglio L, Granieri E, Lauria G. The diagnostic criteria for small fibre neuropathy: from symptoms to neuropathology. Brain. 2008 Jul;131(Pt 7):1912-25. doi: 10.1093/brain/awn093. Epub 2008 Jun 4. PMID 18524793
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Tankisi H, Pugdahl K, Beniczky S, Andersen H, Fuglsang-Frederiksen A. Evidence-based recommendations for examination and diagnostic strategies of polyneuropathy electrodiagnosis. Clin Neurophysiol Pract. 2019 Nov 18;4:214-222. doi: 10.1016/j.cnp.2019.10.005. eCollection 2019. PMID 31886447
- [Background] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Background] Terkawi AS, Abolkhair A, Didier B, Alzhahrani T, Alsohaibani M, Terkawi YS, Almoqbali Y, Tolba YY, Pangililan E, Foula F, Tsang S. Development and validation of Arabic version of the douleur neuropathique 4 questionnaire. Saudi J Anaesth. 2017 May;11(Suppl 1):S31-S39. doi: 10.4103/sja.SJA_97_17. PMID 28616002
- [Background] Eldokla AM, Mohamed-Hussein AA, Fouad AM, Abdelnaser MG, Ali ST, Makhlouf NA, Sayed IG, Makhlouf HA, Shah J, Aiash H. Prevalence and patterns of symptoms of dysautonomia in patients with long-COVID syndrome: A cross-sectional study. Ann Clin Transl Neurol. 2022 Jun;9(6):778-785. doi: 10.1002/acn3.51557. Epub 2022 Apr 8. PMID 35393771
- [Background] Ewing DJ, Martyn CN, Young RJ, Clarke BF. The value of cardiovascular autonomic function tests: 10 years experience in diabetes. Diabetes Care. 1985 Sep-Oct;8(5):491-8. doi: 10.2337/diacare.8.5.491. PMID 4053936
- [Background] Bril V, Perkins BA. Validation of the Toronto Clinical Scoring System for diabetic polyneuropathy. Diabetes Care. 2002 Nov;25(11):2048-52. doi: 10.2337/diacare.25.11.2048. PMID 12401755
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Al Shabasy S, Abbassi M, Finch A, Roudijk B, Baines D, Farid S. The EQ-5D-5L Valuation Study in Egypt. Pharmacoeconomics. 2022 Apr;40(4):433-447. doi: 10.1007/s40273-021-01100-y. Epub 2021 Nov 17. PMID 34786590
- [Background] Bekairy AM, Bustami RT, Almotairi M, Jarab A, Katheri AM, Aldebasi TM, Aburuz S. Validity and reliability of the Arabic version of the the EuroQOL (EQ-5D). A study from Saudi Arabia. Int J Health Sci (Qassim). 2018 Mar-Apr;12(2):16-20. PMID 29599689
- [Background] Vetrugno R, Liguori R, Cortelli P, Montagna P. Sympathetic skin response: basic mechanisms and clinical applications. Clin Auton Res. 2003 Aug;13(4):256-70. doi: 10.1007/s10286-003-0107-5. PMID 12955550
- [Background] Lauria G, Hsieh ST, Johansson O, Kennedy WR, Leger JM, Mellgren SI, Nolano M, Merkies IS, Polydefkis M, Smith AG, Sommer C, Valls-Sole J; European Federation of Neurological Societies; Peripheral Nerve Society. European Federation of Neurological Societies/Peripheral Nerve Society Guideline on the use of skin biopsy in the diagnosis of small fiber neuropathy. Report of a joint task force of the European Federation of Neurological Societies and the Peripheral Nerve Society. Eur J Neurol. 2010 Jul;17(7):903-12, e44-9. doi: 10.1111/j.1468-1331.2010.03023.x. PMID 20642627
- [Background] Telleman JA, Herraets IJ, Goedee HS, van Asseldonk JT, Visser LH. Ultrasound scanning in the diagnosis of peripheral neuropathies. Pract Neurol. 2021 Jun;21(3):186-195. doi: 10.1136/practneurol-2020-002645. Epub 2021 Feb 4. PMID 33541914
- [Background] Tawfik EA, Walker FO, Cartwright MS, El-Hilaly RA. Diagnostic Ultrasound of the Vagus Nerve in Patients with Diabetes. J Neuroimaging. 2017 Nov;27(6):589-593. doi: 10.1111/jon.12452. Epub 2017 May 19. PMID 28524416
- [Background] Ebadi H, Siddiqui H, Ebadi S, Ngo M, Breiner A, Bril V. Peripheral Nerve Ultrasound in Small Fiber Polyneuropathy. Ultrasound Med Biol. 2015 Nov;41(11):2820-6. doi: 10.1016/j.ultrasmedbio.2015.06.011. Epub 2015 Aug 28. PMID 26318562